CLINICAL TRIAL: NCT00432523
Title: An Open, Randomised, Comparative, Multicentre Study of the Immunogenicity and Safety of M-M-R™II Manufactured With Recombinant Human Albumin (rHA) and VARIVAX® When Administered Concomitantly by Intramuscular (IM) Route or Subcutaneous (SC) Route at Two Separate Injection Sites in Healthy Subjects 12 to 18 Months of Age
Brief Title: Immunogenicity and Safety of Concomitant Administration of MMR™ rHA and VARIVAX® by Intramuscular Versus Subcutaneous Route (V205C-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: V205C-011; X04-MMRr-301 (Other: MCMVaccBV (SPMSD) Secondary ID)
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Measles; Mumps; Varicella
Keywords: Prevention of : Measles, Mumps, Rubella and Varicella diseases
MeSH Terms: conditions — Measles; Mumps; Chickenpox; Rubella | interventions — Chickenpox Vaccine

INTERVENTIONS:
Biological: M-M-R™II manufactured with recombinant Human Albumin (rHA) and VARIVAX®

SUMMARY:
Primary objective:

To compare if, when given concomitantly with VARIVAX® by the same route at 12-18 months of age using separate injection sites, a single dose of M-M-RTMII administered by IM route is as immunogenic as a single dose of M-M-RTMII administered by SC route in terms of response rates to measles, mumps and rubella at 42 days following the vaccination.

AND/OR

To compare if, when given concomitantly with M-M-RTMII by the same route at 12-18 months of age using separate injection sites, a single dose of VARIVAX® administered by IM route is as immunogenic as a single dose of VARIVAX® administered by SC route in terms of response rate to varicella at 42 days following the vaccination

Secondary objectives:

* To summarise the antibody titres to measles, mumps, rubella and varicella at 42 days following the vaccination in children immunised with M-M-R™II and VARIVAX® administered concomitantly at two separate injection sites by the same route IM or SC,
* To evaluate the safety profiles of M-M-R™II and VARIVAX® administered concomitantly at two separate injection sites by the same route IM or SC.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject of either gender,
2. Age 12 to 18 months ,
3. Consent form signed by both parent(s) or by the legal representative properly informed about the study,
4. Parent(s) / legal representative able to understand the protocol requirements and to fill in the Diary Card.

Exclusion Criteria:

1. Prior receipt of measles, mumps, rubella or varicella vaccine either alone or in combination vaccine,
2. Known or suspected clinical history of infection with measles, mumps, rubella, varicella or zoster,
3. Any recent (≤30 days) exposure to measles, mumps or rubella,
4. Any recent (≤30 days) exposure to varicella or zoster involving:
5. Any recent (≤3 days) history of febrile illness
6. Any severe chronic disease,
7. Active untreated tuberculosis,
8. Known personal history of seizures,
9. Any known blood dyscrasia, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems,
10. Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection,
11. Any immune impairment or humoral/cellular deficiency, neoplastic disease or depressed
12. Any recent tuberculin test (≤7 days) or scheduled tuberculin test through visit 2,
13. Any previous (≤150 days) receipt of immune serum globulin or any blood-derived products or scheduled to be administered through visit 2,
14. Any recent receipt of an inactivated or a live vaccine (≤30 days) or scheduled vaccination through visit 2

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 752
Dates: Start 2005-01-20 (Actual); Primary Completion 2005-09-05 (Actual); Study Completion 2005-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne FIQUET, MD, Study Director — SPMSD
Locations (2):
- France, France
- Germany, Germany

REFERENCES:
- [Derived] Gillet Y, Habermehl P, Thomas S, Eymin C, Fiquet A. Immunogenicity and safety of concomitant administration of a measles, mumps and rubella vaccine (M-M-RvaxPro) and a varicella vaccine (VARIVAX) by intramuscular or subcutaneous routes at separate injection sites: a randomised clinical trial. BMC Med. 2009 Apr 14;7:16. doi: 10.1186/1741-7015-7-16. PMID 19366435